CLINICAL TRIAL: NCT06891729
Title: Safety and Clinical Validation Study of the Plan A Delivery Lumen Access Device (DLAD)
Brief Title: Plan A Novel Delivery Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Life Sciences (Industry)
Collaborators: Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP100
Record Dates: First submitted 2025-03-08; First posted 2025-03-24 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Male Adults Participants; Vasectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Interventional Arm (Experimental): All participants who provide informed consent and are deemed eligible will be treated with the investigational device immediately prior to their planned vasectomy.
  Interventions: Device: Delivery Lumen Access Device; Device: DLAD

INTERVENTIONS:
Device: Delivery Lumen Access Device — Delivery Lumen Access Device use prior to Vasectomy
Device: DLAD — Participants will be exposed to the DLAD during their planned vasectomy

SUMMARY:
This study will evaluate the safety and usability of the Delivery Lumen Access Device (DLAD) in accessing the vas deferens in up to 30 healthy males. This is a prospective, non-randomized, open label interventional study.

DETAILED DESCRIPTION:
This is a first in human research study, testing an investigational device which is being developed as part of a potential, non-hormonal, long-lasting, reversible male contraceptive system. The device is called the Delivery Lumen Access Device (DLAD) and it is intended to deliver a non-hormonal gel into the vas deferens to block the flow of sperm. Only the DLAD device is being tested in this study; the non-hormonal gel will not be administered. The purpose of this study is to confirm if the DLAD is safe to use and can access the vas deferens. The usability of the DLAD will also be assessed.

Up to 30 men, aged between 18 and 65 years, planning to undergo a vasectomy will be recruited for the study. Following a screening period of up to 30 days, eligible participants will undergo the DLAD procedure during their vasectomy. Post-procedure monitoring and recovery will be performed as per standard of care for a vasectomy procedure.

Participants will be contacted by telephone 14 days after the procedure to check for adverse events and changes in concomitant medications. If the investigator deems it necessary, the 14-day follow-up may be conducted in the clinic. At the investigator's discretion, participants may also be asked to attend unscheduled visits to assess adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject who has already planned to undergo a vasectomy.
2. Male subject who has voluntarily signed and dated the Institutional Review Board (IRB)/Ethics Committee (EC) approved informed consent form (ICF) for this study before initiation of any screening or study-specific procedures.
3. 18 to 65 years of age at the time of consent.
4. Good health for undergoing a vasectomy procedure as confirmed by medical history and physical examination.
5. In the opinion of the Investigator, the subject is suitable to undergo a vasectomy procedure as a form of long-term contraception.

Exclusion Criteria:

1. On exam, has any of the following: one or both vasa not present, abnormal scrotum, large varicocele, hydrocele, filariasis or elephantiasis of scrotum, or an intrascrotal mass that would make the subject not suitable for the study.
2. Prior testicular surgery, testicular injury, or prior vasectomy with vasovasostomy (vasectomy reversal).
3. Has local genital infections such as balanitis, scrotal skin infection, epididymitis, or orchitis, or tender (inflamed) tip of the penis, but may be enrolled after resolution of an acute infection.
4. History of prostatitis or benign prostatic hypertrophy requiring treatment.
5. Has known current coagulopathy or other bleeding disorders.
6. Known allergy to DLAD materials including nickel, stainless steel and silicone.
7. Has cystic fibrosis.
8. Has history of inguinal hernia repair.
9. The subject belongs to a vulnerable population. Vulnerable subject populations are defined as individuals who are incarcerated, handicapped, have cognitive challenges, mental disability, persons in nursing homes, children, impoverished persons, homeless persons, economically or educationally disadvantaged persons, nomads, refugees and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces and persons kept in detention.
10. Currently participating in another study involving an investigational device or drug within the last 30 days prior to the first screening.
11. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.
12. In the opinion of the Investigator, there are issues or concerns that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.
13. Has any condition that, in the opinion of the Investigator, would interfere with evaluation of DLAD product performance or interpretation of patient safety or study results.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Walley, Study Director — Next Life Sciences
Locations (2):
- Epworth HealthCare, Melbourne, Victoria, Australia
- VasectoPro, Québec, Quebec/Canada, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Epworth Healthcare (hospital facility, Australia): Recruitment period from March 20 - April 8, 2025.
  VasectoPro (Medical clinic, Canada): Recruitment period from May 9 - May 25, 2025.
Pre-assignment Details: All enrolled participants were included in the study.
Period: Overall Study
Arm/Group | Interventional Arm
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Arm
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — The mean age was 38.32. The standard deviation was 6.09 and the range was 30.4 to 50.65.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 24
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.32 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 20
  Australia | 4
Physical examination and vital signs. [Count of Participants; unit: Participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Treatment emergent adverse events
Time Frame: 14 days post vasectomy procedure.
Population: TEAES will captured during the procedure and through the 14 day follow up visit and study completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 24
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the first patients screening visit through the last patients Day 14 follow up visit.
Description: Adverse events were captured from the first patients screening visit through the last patients Day 14 follow up visit.
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=24)
Scrotal Pain (Reproductive system and breast disorders) | 4 (4) — Scrotal discomfort
Non Infectious Inflammation (Reproductive system and breast disorders) | 4 (4) — Non-infectious swelling.

LIMITATIONS AND CAVEATS:
Due to the early stage in this clinical program the sample size was relatively small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI's may not publish or discuss the results without consent and review by NLS.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT06891729/Prot_SAP_000.pdf